CLINICAL TRIAL: NCT03142308
Title: Young Surgeons' Satisfaction With the Surgical Training Program in Egyptian University Hospitals: A Multi-center Cross-sectional Study
Brief Title: Surgeons' Satisfaction With the Surgical Training Program in Egypt
Acronym: multi-center
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Collaborators: Cairo University (Other); Ain Shams University (Other); Al-Azhar University (Other); Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed S.A. Shehata, Principle Investigator, Zagazig University
Other Study IDs: 3259/18-122016
Record Dates: First submitted 2017-04-25; First posted 2017-05-05 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Satisfaction
Keywords: Satisfaction; Training program; Egypt; Cross-sectional; Multi-center
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgeons: Young surgeons in all surgical specialities

SUMMARY:
In Egypt, the evidence for quality processes has not been established yet in the current training programs for surgery residents. There are no published articles discussing career satisfaction among surgical residents. Therefore, we are going to conduct a self-designed survey in Egyptian university hospitals to measure residents' satisfaction and display views about their undergraduate surgical education, surgical education during internship year, post-graduate training program, and extracurricular activity during medical school.

ELIGIBILITY:
Inclusion Criteria:

* We will include the Egyptian academic surgeons, within their first 8 years after their graduation. We will include surgeons in general surgery and other surgery subspecialties such as orthopedic surgery, neurosurgery, urology, and plastic surgery

Exclusion Criteria:

* We will exclude surgeons who received part of their training program abroad.

Ages: 26 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents (juniors, sub-seniors, seniors) and assistant lectures in all surgical specialities.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Surgeons' satisfaction with undergraduate surgical education, surgical training during the internship year, and residency using validated questionnaire | Within 8 years of graduation
  By validated questionnaire, we will assess surgeons' satisfaction with lectures, clinical rounds, skill labs during undergraduate, satisfaction with tutorials, operating room, outpatient clinic, ward rounds, and seminars during internship year, satisfaction with theoretical and clinical training program, and number of working hours during the residency.

SECONDARY OUTCOMES:
Define the reasons of dissatisfaction by validated questionnaire. | Within 8 years of graduation
  Using validated questionnaire, we will assess the reasons of dissatisfaction such as insufficient teaching time, dysfunctional curriculum, training environment, and teaching methodology.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No